CLINICAL TRIAL: NCT00978991
Title: Duke Longitudinal Urologic Surgery Patient Outcome Database
Brief Title: Duke Urology Database and Specimen Bank
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Principal Investigator, Judd Moul, Professor of Surgery, Duke University
Other Study IDs: Pro00005140
Record Dates: First submitted 2009-09-15; First posted 2009-09-17 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2013-02

CONDITIONS: Prostate Cancer; Bladder Cancer; Erectile Dysfunction; Incontinence
Keywords: Benign prostate hyperplasia; Erectile dysfunction
MeSH Terms: conditions — Prostatic Neoplasms; Urinary Bladder Neoplasms; Erectile Dysfunction; Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The proposed project is aimed to build a Duke University-specific longitudinal urologic surgery database. It will be used as the main resource to support future research within Urology and Duke University.

DETAILED DESCRIPTION:
Specifically, the database will be used for the following future studies. (i) To characterize the biomarkers/protein signature associated with urological diseases; (ii) To clarify the clinical role of the risk factors and their interactions for early detection and optimized treatment of urological diseases, and improvement of post-treatment quality of life; (iii) To develop algorithms and nomograms to accurately predict the outcome of urological diseases.

Retrospective review of subjects data prior to Institutional Review Board approval and prospective review of data on those consented after Institutional Review Board approval.

ELIGIBILITY:
Inclusion Criteria:

* Duke Urology patients

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Urology
Sampling Method: Non-Probability Sample
Enrollment: 87820 (Actual)
Dates: Start 1988-01; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judd W Moul, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States